CLINICAL TRIAL: NCT04854577
Title: The Postoperative Opioid-Sparing Effect of an Intraoperative Pecto-Intercostal Fascial Block and Opioid-Free Anesthesia in Cardiac Surgery Patients: a Prospective Randomized Controlled Trial
Brief Title: Postoperative Opioid-Sparing Effect of a Pecto-Intercostal Fascial Block and Opioid-Free Anesthesia.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Algemeen Stedelijk Ziekenhuis (Other)
Responsible Party: Principal Investigator, Koen Lapage, M.D., Consultant Anesthesiology, Algemeen Stedelijk Ziekenhuis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APIC2021150303; 2021-002164-43 (EudraCT Number)
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Opioid Free Anaesthesia; Opioid Anaesthesia
Keywords: Analgesics, Opioid; Anesthetics; Central Nervous System Depressants; Dexmedetomidine; Esketamine; Lidocaine; Ropivacaine; Pecto-Intercostal Fascial Plane Block; Physiological Effects of Drugs; Peripheral Nervous System Agents

STUDY DESIGN:
Intervention Model Description: A randomized controlled, outcome assessor blinded study using two parallel study groups
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient will not be made aware of what has been administered. The outcome assessor will be blinded for the group allocation of patients. The investigator, as one of the care providers, nor the care providers can be blinded for the administered anesthetic regimen. The opioid free anesthetic regimen will be conducted by the same anesthesiologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: "Opioid Free Anesthesia with a pecto-intercostal fascial plane block" (Experimental): Patients to whom a standardized opioid free anesthesia consisting of esketamine, lidocaine and dexmedetomidine will be administered with a pre-incisional pecto-intercostal fascial plane block.
  Interventions: Procedure: Opioid Free Anesthesia
- Control group: "Traditional Opioid-based Anesthetic Regimen" (Active Comparator): Patients who will receive a traditional opioid based anesthetic regimen. The administered dose of opioids is at the discretion of the attending anesthesiologist.
  Interventions: Procedure: Traditional Anesthetic Regimen

INTERVENTIONS:
Procedure: Opioid Free Anesthesia — Patients will be administered a combination of a pre-incisional pecto-intercostal fascial plane block and a standardized opioid free anesthetic regimen consisting of dexmedetomidine, esketamine and lidocaine.
  Arms: Intervention group: "Opioid Free Anesthesia with a pecto-intercostal fascial plane block"
Procedure: Traditional Anesthetic Regimen — Patients will be administered a traditional anesthetic regimen which is based on sufentanil dosage. The dosage is at the discretion of the attending anesthesiologist.
  Arms: Control group: "Traditional Opioid-based Anesthetic Regimen"

SUMMARY:
The present study aims to assess the difference in postoperative opioid consumption between patients who intraoperatively receive a pecto-intercostal facial block combined with opioid-free anesthesia versus a traditional opioid-based regimen for cardiac surgery. The literature on opioid-free anesthesia for cardiac surgery is minimal and solely consists of case reports and retrospective studies. Nevertheless, these reports show the feasibility of opioid-free anesthesia. The purpose of this study is to assess the opioid-sparing effect and efficacy of combining an opioid-free anesthetic regimen with a pecto-intercostal fascial plane block (PIFB) in patients undergoing cardiac surgery.

We hypothesize that opioid-free cardiac anesthesia with an intraoperative PIFB significantly reduces postoperative opioid consumption in comparison to a high-dose opioid intraoperative regimen.

DETAILED DESCRIPTION:
Patients, aged 18 years or older, scheduled for coronary artery bypass graft surgery (CABG) with a complete midline sternotomy as surgical approach will be recruited for this study.

Patients planned for this particular surgical procedure will be recruited and allocated to one of 2 groups:

1. "Intervention" group: Opioid-free anesthetic regimen with a pre-incisional pecto-intercostal fascial plane block (PIFB);
2. "Control" group: traditional opiate-based anesthetic regimen in which the dosage of the opioids is at the discretion of the attending anesthesiologist.

Based on our power analysis, each group will consist of 64 patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Patients scheduled for coronary artery bypass graft surgery (CABG), which includes a complete midline sternotomy.

Exclusion Criteria:

* CABG surgery which did not include a complete midline sternotomy
* Valve surgery
* Aortic surgery
* Emergency cardiac surgery
* Known allergy for ropivacaine
* Participation in another clinical trial
* Known drug abuse
* Preoperative cognitive dysfunction
* Preoperative pain therapy with opioids or anticonvulsants 14 days before surgery
* Patients unable to use Patient Controlled Analgesia (PCA)
* Need of reintubation after initial extubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Postoperative morphine consumption | Day 2
  The total amount of morphine used postoperatively in the intensive care unit until discharge.

SECONDARY OUTCOMES:
Time until extubation | Day 0
  The time between ICU-arrival and extubation
Mean visual analogue score (VAS) pain score at rest | Day 2
  The mean VAS pain score at rest at 24 hours and 48 hours after extubation.
Mean visual analogue score (VAS) pain score whilst coughing | Day 2
  The mean VAS pain score whilst coughing at 24 hours and 48 hours after extubation.
Incidence of postoperative nausea and vomiting | Day 2
  Incidence of postoperative nausea and vomiting (PONV)
Incidence of postoperative delirium | Day 2
  Incidence of postoperative delirium using the Confusion Assessment Method for ICU
Mean length of ICU stay | Day 2
  The mean length of ICU stay, reported in hours.

CONTACTS AND LOCATIONS:
Overall Officials: Koen Lapage, M.D., Principal Investigator — Department of Anesthesiology, Pain and Intensive Care Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwanten LE, O'Brien B, Anwar S. Opioid-Based Anesthesia and Analgesia for Adult Cardiac Surgery: History and Narrative Review of the Literature. J Cardiothorac Vasc Anesth. 2019 Mar;33(3):808-816. doi: 10.1053/j.jvca.2018.05.053. Epub 2018 Jun 5. PMID 30064852
- [Background] Bignami E, Castella A, Pota V, Saglietti F, Scognamiglio A, Trumello C, Pace MC, Allegri M. Perioperative pain management in cardiac surgery: a systematic review. Minerva Anestesiol. 2018 Apr;84(4):488-503. doi: 10.23736/S0375-9393.17.12142-5. Epub 2017 Oct 12. PMID 29027773
- [Background] Wheeler M, Oderda GM, Ashburn MA, Lipman AG. Adverse events associated with postoperative opioid analgesia: a systematic review. J Pain. 2002 Jun;3(3):159-80. doi: 10.1054/jpai.2002.123652. No abstract available. PMID 14622770
- [Background] Ochroch J, Usman A, Kiefer J, Pulton D, Shah R, Grosh T, Patel S, Vernick W, Gutsche JT, Raiten J. Reducing Opioid Use in Patients Undergoing Cardiac Surgery - Preoperative, Intraoperative, and Critical Care Strategies. J Cardiothorac Vasc Anesth. 2021 Jul;35(7):2155-2165. doi: 10.1053/j.jvca.2020.09.103. Epub 2020 Sep 15. PMID 33069556
- [Background] Kessler ER, Shah M, Gruschkus SK, Raju A. Cost and quality implications of opioid-based postsurgical pain control using administrative claims data from a large health system: opioid-related adverse events and their impact on clinical and economic outcomes. Pharmacotherapy. 2013 Apr;33(4):383-91. doi: 10.1002/phar.1223. PMID 23553809
- [Background] Hagemeier NE. Introduction to the opioid epidemic: the economic burden on the healthcare system and impact on quality of life. Am J Manag Care. 2018 May;24(10 Suppl):S200-S206. PMID 29851449
- [Background] Shipton EA, Shipton EE, Shipton AJ. A Review of the Opioid Epidemic: What Do We Do About It? Pain Ther. 2018 Jun;7(1):23-36. doi: 10.1007/s40122-018-0096-7. Epub 2018 Apr 6. PMID 29623667
- [Background] Brat GA, Agniel D, Beam A, Yorkgitis B, Bicket M, Homer M, Fox KP, Knecht DB, McMahill-Walraven CN, Palmer N, Kohane I. Postsurgical prescriptions for opioid naive patients and association with overdose and misuse: retrospective cohort study. BMJ. 2018 Jan 17;360:j5790. doi: 10.1136/bmj.j5790. PMID 29343479
- [Background] Clarke H, Soneji N, Ko DT, Yun L, Wijeysundera DN. Rates and risk factors for prolonged opioid use after major surgery: population based cohort study. BMJ. 2014 Feb 11;348:g1251. doi: 10.1136/bmj.g1251. PMID 24519537
- [Background] Cardinale JP, Gilly G. Opiate-Free Tricuspid Valve Replacement: Case Report. Semin Cardiothorac Vasc Anesth. 2018 Dec;22(4):407-413. doi: 10.1177/1089253218771342. Epub 2018 Apr 20. PMID 29676223
- [Background] Chanowski EJP, Horn JL, Boyd JH, Tsui BCH, Brodt JL. Opioid-Free Ultra-Fast-Track On-Pump Coronary Artery Bypass Grafting Using Erector Spinae Plane Catheters. J Cardiothorac Vasc Anesth. 2019 Jul;33(7):1988-1990. doi: 10.1053/j.jvca.2018.10.012. Epub 2018 Oct 13. No abstract available. PMID 30424939
- [Background] Guinot PG, Spitz A, Berthoud V, Ellouze O, Missaoui A, Constandache T, Grosjean S, Radhouani M, Anciaux JB, Parthiot JP, Merle JP, Nowobilski N, Nguyen M, Bouhemad B. Effect of opioid-free anaesthesia on post-operative period in cardiac surgery: a retrospective matched case-control study. BMC Anesthesiol. 2019 Jul 31;19(1):136. doi: 10.1186/s12871-019-0802-y. PMID 31366330
- [Background] Caruso TJ, Lawrence K, Tsui BCH. Regional anesthesia for cardiac surgery. Curr Opin Anaesthesiol. 2019 Oct;32(5):674-682. doi: 10.1097/ACO.0000000000000769. PMID 31356362
- [Background] Landoni G, Isella F, Greco M, Zangrillo A, Royse CF. Benefits and risks of epidural analgesia in cardiac surgery. Br J Anaesth. 2015 Jul;115(1):25-32. doi: 10.1093/bja/aev201. PMID 26089444
- [Background] Smith LM, Barrington MJ; St Vincent's Hospital, Melbourne. Ultrasound-guided blocks for cardiovascular surgery: which block for which patient? Curr Opin Anaesthesiol. 2020 Feb;33(1):64-70. doi: 10.1097/ACO.0000000000000818. PMID 31833864
- [Background] Khera T, Murugappan KR, Leibowitz A, Bareli N, Shankar P, Gilleland S, Wilson K, Oren-Grinberg A, Novack V, Venkatachalam S, Rangasamy V, Subramaniam B. Ultrasound-Guided Pecto-Intercostal Fascial Block for Postoperative Pain Management in Cardiac Surgery: A Prospective, Randomized, Placebo-Controlled Trial. J Cardiothorac Vasc Anesth. 2021 Mar;35(3):896-903. doi: 10.1053/j.jvca.2020.07.058. Epub 2020 Jul 24. PMID 32798172
- [Background] Kumar AK, Chauhan S, Bhoi D, Kaushal B. Pectointercostal Fascial Block (PIFB) as a Novel Technique for Postoperative Pain Management in Patients Undergoing Cardiac Surgery. J Cardiothorac Vasc Anesth. 2021 Jan;35(1):116-122. doi: 10.1053/j.jvca.2020.07.074. Epub 2020 Jul 30. PMID 32859487
- [Background] Chan JL, Miller JG, Murphy M, Greenberg A, Iraola M, Horvath KA. A Multidisciplinary Protocol-Driven Approach to Improve Extubation Times After Cardiac Surgery. Ann Thorac Surg. 2018 Jun;105(6):1684-1690. doi: 10.1016/j.athoracsur.2018.02.008. Epub 2018 Mar 9. PMID 29530778
- [Background] Berthoud V, Ellouze O, Nguyen M, Konstantinou M, Aho S, Malapert G, Girard C, Guinot PG, Bouchot O, Bouhemad B. Serratus anterior plane block for minimal invasive heart surgery. BMC Anesthesiol. 2018 Oct 20;18(1):144. doi: 10.1186/s12871-018-0614-5. PMID 30340525